CLINICAL TRIAL: NCT04310098
Title: Cerebral Autosomal Dominant Arteriopathy With Subcortical Infarcts and Leukoencephalopathy Registry Study
Brief Title: CADASIL Registry Study
Status: Recruiting | Type: Observational
Sponsor: Bin Cai (Other)
Responsible Party: Sponsor-Investigator, Bin Cai, Professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH of FMU [2019]244-1
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cadasil
MeSH Terms: conditions — CADASIL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CADASIL patients
- Asymptomatic carriers of CADASIL
- Relatives of CADASIL patients and carriers
- Unrelated healthy controls

SUMMARY:
The aim of this study is to determine the clinical spectrum and natural progression of Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leukoencephalopathy (CADASIL) and related disorders in a prospective multicenter study, to assess the clinical, genetic and epigenetic features of patients with CADASIL , to optimize clinical management.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent.
2. Age>18
3. Clinical diagnosis of patients with CADASIL,and confirmed by genetic test or skin biopsy
4. Asymptomatic NOTCH3 mutation carriers
5. Relatives of CADASIL patients or carriers
6. Unrelated healthy controls

Exclusion Criteria:

1. Unable to cooperate with inspectors
2. Serious systemic illness, such as heart, liver, kidney disease or major mental illness
3. Contraindications for imaging examination

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed in hosipital and their's family
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2039-03-09 (Estimated); Study Completion 2049-03-09 (Estimated)

PRIMARY OUTCOMES:
Overall outcomes in CADASIL patients | From date of enrollment until the date of death from any cause, assessed up to 20years
  record the occurrence of stroke and use modified Rankin Scale (mRS) to measure the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.

SECONDARY OUTCOMES:
The correlation of genotype and phenotype | From date of enrollment until the date of death from any cause, assessed up to 20years
  Genotype is defined by NOTCH3 pathogenic variant position and phenotype is defined by clinical types and characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology , First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian, China